CLINICAL TRIAL: NCT02828904
Title: Retrospective Cohort Study on the RIsk of VEnous Thromboembolism Associated With the Use of Combined Oral Contraceptives Containing Chlormadinone Acetate/Ethinylestradiol and Levonorgestrel/Ethinylestradiol
Brief Title: RIVET - Retrospective Cohort Study on the Risk of Venous Thromboembolism
Acronym: RIVET-RCS
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Responsible Party: Principal Investigator, Klaas Heinemann, MD, PhD, PhD, MD, MSc, MBA, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2014_05
Record Dates: First submitted 2016-06-20; First posted 2016-07-12 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Users of Chlormadinone Acetate (CMA) combined with Ethinylestradiol (EE): CMA/EE users are defined as
  * aged 15 to 49 years
  * Participation in one of the 4 observational studies conducted between 2000 and 2019 (LASS/EURAS-OC, INAS-OC, INAS-SCORE, INAS-FOCUS)
  * COC new user (starters, switchers, and re-starters)
- Users of Levonorgestrel (LNG) combined with Ethinylestradiol (EE): LNG/EE users are defined as
  * aged 15 to 49 years
  * Participation in one of the 4 observational studies conducted between 2000 and 2019 (LASS/EURAS-OC, INAS-OC, INAS-SCORE, INAS-FOCUS)
  * COC new user (starters, switchers, and re-starters)

SUMMARY:
The risk of venous thromboembolism (VTE) associated with the use of chlormadinone acetate (CMA) compared to the gold-standard progestin levonorgestrel (LNG) as component of combined oral contraceptives (COC) is currently unknown. The Pharmacovigilance Risk Assessment Committee (PRAC) of the European Medicines Agency (EMA) recommended a pooled analysis of four prospective cohort studies carried out by the Berlin Center for Epidemiology and Health Research (ZEG Berlin) in order to clarify whether CMA-containing COCs carry a different VTE risk compared to LNG-containing COCs.

DETAILED DESCRIPTION:
This study is designed as a retrospective cohort study. ZEG Berlin conducted several large prospective cohort studies on the risk of VTE associated with the use of hormonal contraceptives. Four of these studies included a substantial number of women using CMA/EE or LNG/EE-containing COCs. For this study, the data on CMA/EE and LNG/EE from the following four prospective cohort studies are combined: 1) EURAS-OC/LASS 2) INAS-OC 3) INAS-SCORE and 4) INAS-FOCUS.

Participants will be identified retrospectively from a pooled dataset which comprises four large, controlled, prospective, non-interventional active surveillance studies that focused on the risk of VTE associated with the use of combined oral contraceptives. All data were prospectively collected by ZEG Berlin and follow the EURAS/INAS study design. Inclusion and exclusion criteria, the method of patient recruitment and follow-up as well as research methods were similar across studies.

The EURAS-OC/LASS study was conducted in Europe only; the other three studies are transatlantic studies that include subjects from both Europe and the United States of America.

This analysis is specifically designed to assess the risk of VTE associated with the use of COCs containing CMA/EE compared to LNG/EE.

ELIGIBILITY:
Inclusion: female, aged 15 to 49 years, participation in one of the 4 observational studies conducted between 2000 and 2019 (LASS/EURAS-OC, INAS-OC, INAS-SCORE, INAS-FOCUS), COC new user (starters, switchers, and re-starters), applied COCs: CMA/EE or LNG/EE.

Exclusion of women with a personal history of VTE.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be identified retrospectively from a pooled dataset which comprises four large, controlled, prospective, non-interventional active surveillance studies that focused on the risk of VTE associated with the use of combined oral contraceptives. All data were prospectively collected by ZEG Berlin and follow the EURAS/INAS study design. Inclusion and exclusion criteria, the method of patient recruitment and follow-up as well as research methods were similar across studies.
Sampling Method: Probability Sample
Enrollment: 124000 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
The risk of venous thromboembolic events (VTE) in the cohort of users of combined oral contraceptives (COCs) containing 2 mg CMA/30 µg EE compared to 0.15 mg LNG/30 µg EE. | VTEs will be identified during the follow-up intervals, typically scheduled every 6 - 12 months, with a maximum follow-up of 10 years.
  VTE risk of users of CMA 2mg / EE 30µg compared to the VTE risk of users of LNG 0.15 mg / EE 30µg.

SECONDARY OUTCOMES:
To assess the risk of venous thromboembolic events stratified by: COC user type, age and BMI | During the follow-up intervals, typically scheduled every 6 - 12 months, with a maximum follow-up of 10 years.
To assess the risk of VTE in the sub-cohort of users of COCs containing CMA compared to LNG both combined with ≤30 µg EE. | During the follow-up intervals, typically scheduled every 6 - 12 months, with a maximum follow-up of 10 years.
To characterize the baseline risk of users of the two formulations (lifetime history of co-morbidity, prognostic factors for VTE, co-medication, socio-demographic and life¬style data). | During the follow-up intervals, typically scheduled every 6 - 12 months, with a maximum follow-up of 10 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Epidemiology and Health Research Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No